CLINICAL TRIAL: NCT05096702
Title: Operational Feasibility of Appropriate Radical Cure of Plasmodium Vivax With Tafenoquine or Primaquine After Quantitative G6PD Testing in Brazil
Acronym: Trust
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fundação de Medicina Tropical Dr. Heitor Vieira Dourado (Other)
Collaborators: Centro de Pesquisa em Medicina Tropical (Unknown); Medicines for Malaria Venture (Other); Ministry of Health, Brazil (Other Government); Secretária Municipal de Saúde de Manaus (Unknown); Secretária Estadual de Saúde do Amazonas (Unknown)
Responsible Party: Sponsor
Other Study IDs: CAAE: 16867319.6.0000.0008
Record Dates: First submitted 2021-09-27; First posted 2021-10-27 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Malaria, Vivax; G6PD Deficiency
Keywords: G6PD deficiency; tafenoquine; primaquine; G6PD screening; Operational study; Brazil
MeSH Terms: conditions — Malaria, Vivax; Glucosephosphate Dehydrogenase Deficiency | interventions — tafenoquine; Primaquine

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Tafenoquine (TQ): Patients aged ≥16 years, G6PD activity ≥ 6.1 IU/gHb, not pregnant or breastfeeding, will receive single-dose TQ in addition to standard blood schizonticidal drug.
  Interventions: Drug: Tafenoquine
- Daily primaquine (PQ) for 7 days: Patients aged ≥ 6 months, with G6PD activity between 4.1 and 6.0 IU/gHb, not pregnant or breastfeeding for < 1 month, will receive daily PQ in addition to standard blood schizonticidal drug.
  Interventions: Drug: Primaquine
- Weekly primaquine for 8 weeks: Patients aged ≥ 6 months, with G6PD activity ≤ 4.0 IU/gHb, not pregnant or breastfeeding for < 1 month, will receive weekly once-a-week PQ for eight weeks in addition to standard blood schizonticidal drug.
  Interventions: Drug: Primaquine

INTERVENTIONS:
Drug: Tafenoquine — Tafenoquine 300 mg (2x150mg tablets)
  Other Names: Kozenis
  Groups: Tafenoquine (TQ)
Drug: Primaquine — Daily primaquine adjusted by weight (0.5 mg/kg/day for 7 days)
  Groups: Daily primaquine (PQ) for 7 days
Drug: Primaquine — Weekly primaquine adjusted by weight (0.75mg/kg/week for 8 weeks)
  Groups: Weekly primaquine for 8 weeks

SUMMARY:
This is an observational study carried out in Brazil in patients with P. vivax malaria. The study will be carried out in the municipalities of Manaus (state of Amazonas) and Porto Velho (state of Rondônia).

G6PD and TQ tests will be provided to health facilities by municipal health authorities using the common route for the provision of drugs and diagnostics. PQ and other antimalarial drugs are already available in Brazil.

Designated personnel at the health facilities will be trained to perform the G6PD quantitative test procedure and the radical healing treatment algorithm by the Lead Researcher (RP) team and municipal authorities using teaching materials developed by the sponsors.

The study design is based on the secondary use of data routinely collected from all malaria patients in the Epidemiological Surveillance Information System for Malaria (SIVEP-Malaria) by the Ministry of Health (MS). Data from all malaria patients are routinely collected through SIVEP forms by health professionals (HP) and entered into the SIVEP database by the municipality staff.

The SIVEP form will be adapted by the MS to collect information about the G6PD test, TQ treatment and signs of hemolysis. The retrospective data from all patients will be entered into a new database by the municipality staff during the study period and the relevant data will be automatically exported weekly to the SIVEP database. The study team will only have access to unidentified data, according to the access levels that will be assigned to each member in the system. Only the municipality's team will have access to the identified patient data. In addition to the data collected on the SIVEP forms, the PR team will ask the two referral hospitals that routinely receive all admissions due to AHA to perform a regular screening of electronic hospital admission records for patients with signs of AHA (renal failure, jaundice, blood transfusion, malaria). All identified cases will be investigated using hospital records and SIVEP forms. Confirmed information about drug-induced AHA will be linked to the patient record recorded in the database. The PR team will also contribute to pharmacovigilance training. Physicians at tertiary-level health units will report side effects through the VigiMed system, from the National Health Surveillance Agency (ANVISA).Finally, the additional costs of implementing the G6PD and TQ tests will be collected along with the study at the health facilities.

Since the study is based on retrospective data collection, and the adoption of TQ and G6PD testing will be done by the municipality, the G6PD testing and the treatment of patients with TQ or PQ will be carried out in accordance with the treatment policy , that is, regardless of the study.

The study will be carried out in phases:

- 1st phase (approximately 3 months): Training and provision of G6PD and TQ tests will initially be limited to 10 high-complexity and intermediate-complexity units (referral hospitals, hospitals, emergency care units, polyclinics). Data will be collected from patients with P. vivax treated at these health facilities.

An interim analysis will be performed after collecting data from 600 patients with P. vivax ≥ 16 years, who have not been treated for vivax malaria in the past 60 days, in the study database in order to decide whether the study can be extended to less complex health units. The decision will be made by an Independent Study Oversight Committee (ISOC).

If the interim results of Phase 1 are found to be unsatisfactory, ISOC may decide not to extend the study to primary care units until improvements in the educational program are implemented and/or additional support is provided to health professionals. Additional interim analyzes will be performed as appropriate.

- 2nd phase (approximately 9 months) [CURRENT PHASE]: if approved by ISOC, the study will be extended to less complex health units (basic health units, family health units and other primary care services) and other high and medium complexity of health in the selected municipalities. After staff training, G6PD and TQ testing will be provided to these health facilities by municipal health authorities.

During this 2nd phase, data will continue to be collected from patients with P. vivax treated by the 1st phase tertiary care units.

- An additional interim analysis will be performed after data from 600 patients with P. vivax ≥16 years old, who have not been treated for P. vivax malaria in the past 60 days, from primary care units are collected in the study database ( approximately 3 months after the start of the 2nd phase).

The study will continue while the interim analyzes are being carried out. Final results will be analyzed and validated by ISOC. The study is expected to take approximately 15 months.

DETAILED DESCRIPTION:
This is an observational study carried out in Brazil in patients with P. vivax malaria. The study will be carried out in the municipalities of Manaus (state of Amazonas) and Porto Velho (state of Rondônia).

G6PD and TQ tests will be provided to health facilities by municipal health authorities using the common route for the provision of drugs and diagnostics. PQ and other antimalarial drugs are already available in Brazil.

Designated personnel at the health facilities will be trained to perform the G6PD quantitative test procedure and the radical healing treatment algorithm by the Lead Researcher (RP) team and municipal authorities using teaching materials developed by the sponsors.

The study design is based on the secondary use of data routinely collected from all malaria patients in the Epidemiological Surveillance Information System for Malaria (SIVEP-Malaria) by the Ministry of Health (MS). Data from all malaria patients are routinely collected through SIVEP forms by health professionals (HP) and entered into the SIVEP database by the municipality staff.

The SIVEP form will be adapted by the MS to collect information about the G6PD test, TQ treatment and signs of hemolysis. The retrospective data from all patients will be entered into a new database by the municipality staff during the study period and the relevant data will be automatically exported weekly to the SIVEP database. The study team will only have access to unidentified data, according to the access levels that will be assigned to each member in the system. Only the municipality's team will have access to the identified patient data. In addition to the data collected on the SIVEP forms, the PR team will ask the two referral hospitals that routinely receive all admissions due to AHA to perform a regular screening of electronic hospital admission records for patients with signs of AHA (renal failure, jaundice, blood transfusion, malaria). All identified cases will be investigated using hospital records and SIVEP forms. Confirmed information about drug-induced AHA will be linked to the patient record recorded in the database. The PR team will also contribute to pharmacovigilance training. Physicians at tertiary-level health units will report side effects through the VigiMed system, from the National Health Surveillance Agency (ANVISA).Finally, the additional costs of implementing the G6PD and TQ tests will be collected along with the study at the health facilities.

Since the study is based on retrospective data collection, and the adoption of TQ and G6PD testing will be done by the municipality, the G6PD testing and the treatment of patients with TQ or PQ will be carried out in accordance with the treatment policy , that is, regardless of the study.

The study will be carried out in phases:

- 1st phase (approximately 3 months): Training and provision of G6PD and TQ tests will initially be limited to 10 high-complexity and intermediate-complexity units (referral hospitals, hospitals, emergency care units, polyclinics). Data will be collected from patients with P. vivax treated at these health facilities.

An interim analysis will be performed after collecting data from 600 patients with P. vivax ≥ 16 years, who have not been treated for vivax malaria in the past 60 days, in the study database in order to decide whether the study can be extended to less complex health units. The decision will be made by an Independent Study Oversight Committee (ISOC).

If the interim results of Phase 1 are found to be unsatisfactory, ISOC may decide not to extend the study to primary care units until improvements in the educational program are implemented and/or additional support is provided to health professionals. Additional interim analyzes will be performed as appropriate.

- 2nd phase (approximately 9 months) [CURRENT PHASE]: if approved by ISOC, the study will be extended to less complex health units (basic health units, family health units and other primary care services) and other high and medium complexity of health in the selected municipalities. After staff training, G6PD and TQ testing will be provided to these health facilities by municipal health authorities.

During this 2nd phase, data will continue to be collected from patients with P. vivax treated by the 1st phase tertiary care units.

- An additional interim analysis will be performed after data from 600 patients with P. vivax ≥16 years old, who have not been treated for P. vivax malaria in the past 60 days, from primary care units are collected in the study database ( approximately 3 months after the start of the 2nd phase).

The study will continue while the interim analyzes are being carried out. Final results will be analyzed and validated by ISOC. The study is expected to take approximately 15 months.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of P. vivax malaria (parasitologically confirmed by microscopy or rapid diagnostic test) over six months of age.

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will be carried out in Brazil, in the municipalities of Manaus (state of Amazonas) and Porto Velho (state of Rondônia).Relevant staff members at health facilities will be trained by RP staff and municipal authorities using educational material on the need and use of G6PD testing, treatment algorithm based on G6PD activity levels, TQ adverse events and PQ, identifying, reporting and managing adverse events to ANVISA and MS (completion of the SIVEP DEMO form).
Sampling Method: Probability Sample
Enrollment: 16000 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2023-09-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of P. vivax patients ≥16 years of age treated or not with TQ according to the appropriate level of G6PD enzyme activity. | After the inclusion of 600 patients, approximately 15 months after study start.

SECONDARY OUTCOMES:
Percentage of patients with P. vivax ≥6 months treated or not with PQ according to the appropriate level of G6PD enzyme activity | 15 months after study start
Description of the characteristics of patients treated with TQ or PQ | 15 months after study start
Frequency of drug-induced acute hemolytic anemia (AHA) | 15 months after study start
  Proportion of participants that reported signs and symptoms of hemolysis after P. vivax treatment on malaria notification forms
Hospitalization due to confirmed drug-induced AHA | 15 months after study start
  Proportion of participants hospitalized due drug-induced AHA after malaria treatment, screened in electronic medical records at local reference units and the national hospitalization database.

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Lacerda, MD, PhD, Principal Investigator — Fundação de Medicina Tropical Dr. Heitor Vieira Dourado; Dhelio Batista, MD, PhD, Principal Investigator — Centro de Pesquisa em Medicina Tropical (CEPEM)
Locations (41):
- Brazil (41):
  - Fundação de Medicina Tropical Dr Heitor Vieira Dourado, Manaus, Amazonas
  - Bela Vista, Manaus, Amazonas
  - Campos Salles (Base), Manaus, Amazonas
  - Colônia Antônio Aleixo, Manaus, Amazonas
  - Cooperativa I, Manaus, Amazonas
  - Cueiras (UBSR), Manaus, Amazonas
  - Efigênio Salles (UBSR), Manaus, Amazonas
  - Grande Vitória, Manaus, Amazonas
  - João Paulo II, Manaus, Amazonas
  - Pau Rosa (UBSR), Manaus, Amazonas
  - Platão Araújo (Base), Manaus, Amazonas
  - Santa Inês, Manaus, Amazonas
  - São Pedro (UBSR), Manaus, Amazonas
  - União da Vitória, Manaus, Amazonas
  - Centro de Pesquisa em Medicina Tropical (Cepem), Porto Velho, Rondônia
  - UBS Abunã, Porto Velho, Rondônia
  - UBS Agrovila, Porto Velho, Rondônia
  - UBS Calama, Porto Velho, Rondônia
  - UBS Calderita, Porto Velho, Rondônia
  - UBS Cujubim, Porto Velho, Rondônia
  - UBS Extrema, Porto Velho, Rondônia
  - UBS Fortaleza do Abunã, Porto Velho, Rondônia
  - UBS Jacy-Paraná, Porto Velho, Rondônia
  - UBS José Adelino, Porto Velho, Rondônia
  - UBS Nazaré, Porto Velho, Rondônia
  - UBS Nova Califórnia, Porto Velho, Rondônia
  - UBS Nova Mutum, Porto Velho, Rondônia
  - UBS Palmares, Porto Velho, Rondônia
  - UBS Rio das Garças, Porto Velho, Rondônia
  - UBS Rio Pardo, Porto Velho, Rondônia
  - UBS Ronaldo Aragão, Porto Velho, Rondônia
  - UBS São Carlos, Porto Velho, Rondônia
  - UBS União Bandeirantes, Porto Velho, Rondônia
  - UBS Vila DNIT, Porto Velho, Rondônia
  - UBS Vista Alegre, Porto Velho, Rondônia
  - Upa Zona Leste, Porto Velho, Rondônia
  - SPA Hospital Chapot Prevost, Manaus
  - Upa Campos Sales, Manaus
  - UPA Danilo Corrêa, Manaus
  - UPA José Rodrigues, Manaus
  - Policlínica Ana Adelaide, Rondônia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brito M, Rufatto R, Brito-Sousa JD, Murta F, Sampaio V, Balieiro P, Baia-Silva D, Castro V, Alves B, Alencar A, Duparc S, Grewal Daumerie P, Borghini-Fuhrer I, Jambert E, Peterka C, Edilson Lima F Jr, Carvalho Maia L, Lucena Cruz C, Maciele B, Vasconcelos M, Machado M, Augusto Figueira E, Alcirley Balieiro A, Batista Pereira D, Lacerda M. Operational effectiveness of tafenoquine and primaquine for the prevention of Plasmodium vivax recurrence in Brazil: a retrospective observational study. Lancet Infect Dis. 2024 Jun;24(6):629-638. doi: 10.1016/S1473-3099(24)00074-4. Epub 2024 Mar 4. PMID 38452779
- [Derived] Brito M, Rufatto R, Murta F, Sampaio V, Balieiro P, Baia-Silva D, Castro V, Alves B, Alencar A, Duparc S, Grewal Daumerie P, Borghini-Fuhrer I, Jambert E, Peterka C, Edilson Lima F Jr, Carvalho Maia L, Lucena Cruz C, Maciele B, Vasconcelos M, Machado M, Augusto Figueira E, Alcirley Balieiro A, Menezes A, Ataides R, Batista Pereira D, Lacerda M. Operational feasibility of Plasmodium vivax radical cure with tafenoquine or primaquine following point-of-care, quantitative glucose-6-phosphate dehydrogenase testing in the Brazilian Amazon: a real-life retrospective analysis. Lancet Glob Health. 2024 Mar;12(3):e467-e477. doi: 10.1016/S2214-109X(23)00542-9. PMID 38365417